CLINICAL TRIAL: NCT01798381
Title: The Relationship of Essential Fatty Acids to Cognitive, Electrophysiological and Behavioural Function in Adults With Attention Deficit Hyperactivity Disorder and Controls
Brief Title: Essential Fatty Acids in Adult ADHD
Acronym: OCEAN-GER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Michael Rösler, Prof. Dr., Universität des Saarlandes
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OCEAN-GER
Record Dates: First submitted 2013-02-19; First posted 2013-02-25 (Estimated); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Adult Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Fatty Acids, Essential

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Essential fatty acids (Active Comparator): Omega-3
  Interventions: Dietary Supplement: Essential fatty acids
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Dietary Supplement: Essential fatty acids

INTERVENTIONS:
Dietary Supplement: Essential fatty acids

SUMMARY:
The aim of this project is to investigate the effect of a dietary supplementation with essential fatty acids in adults on cognitive functions related to attention and impulse control in the general population and in individuals with a diagnosis of attention deficit hyperactivity disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV ADHD

Exclusion Criteria:

* any acute psychiatric disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Wender Reimherr Adult Attention Deficit Disorder Scale (WRAADDS) | 6 months
  Psychopatholoy of adult ADHD

SECONDARY OUTCOMES:
Short and long interval cortical inhibition (SICI and LICI) | 6 months
  Motoric evoced potentials by transcranial magnetic stimulation (TMS)

OTHER OUTCOMES:
Cued continous performance test - QB-version | 6 months
  Motorhyper activity, concentration and impulsivity in adult ADHD patients

CONTACTS AND LOCATIONS:
Locations (1):
- Saarland University Hospital, Homburg/Saar, Saarland, Germany